CLINICAL TRIAL: NCT03576300
Title: Comparison of Ocular Surface Features in Patients With Diabetes and Dry Eye Syndrome
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Hong Qi, MD.PHD., Peking University Third Hospital
Other Study IDs: IRB00006761-M2017354
Record Dates: First submitted 2018-06-11; First posted 2018-07-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Dry Eye Syndrome; Diabetes Mellitus Type 2
Keywords: ocular surface
MeSH Terms: conditions — Dry Eye Syndromes; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tears from the subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (4):
- control: subjects without dry eye and diabetes
- patients with diabetes and dry eye: diabetic patients with dry eye
- diabetics without dry eye syndrome: diabetic patients without dry eye
- dry eye syndrome patients without diabetes: non-diabetic patients with dry eye

SUMMARY:
The study aims to compare the differences of ocular surface features in controls and patients with diabetes and dry eye syndrome, to thoroughly evaluate the ocular surface health of diabetics, and to find out the relationship between dry eye syndrome and diabetes

DETAILED DESCRIPTION:
In this study, we perform a completely comparison of ocular surface characteristic including the Ocular Surface Disease Index (OSDI) questionnaire,tearfilm break up time(BUT),corneal fluorescein scores(CFS),Shirmer test,corneal sensitivity)among diabetic patients with DE, diabetic patients without DE, non-diabetic patients with DE and normal subjects and analysis of EGF, IL-17A, IL-1β, IL-8 and TNF-α in tears and their clinical correlations are also performed to investigate potential biomarkers for diagnosis of diabetic with DE.

ELIGIBILITY:
Inclusion Criteria:

1. dry eye diagnosis according to Expert's Consensus About Clinical Diagnosis and Treatment（Corneal Disease Group of Ophthalmological Society, Chinese Medical Association）: ①OSDI≥13，②positive dry eye soigns(ST≤10mm/5min；BUT≤10s；CFS>0)
2. type 2 diabetes diagnosis according to American Diabetes Association：Standards of Medical Care in Diabetes -2017(ADA, American Diabetes Association)
3. Willing to sign the consent form.

Exclusion Criteria:

1. Having known Eye infection, allergy, malformation, abnormal eye movement
2. Exclusion of eye injury, any kind of eye surgery
3. Exclusion of other disease may cause neuropathy or influence tear producing
4. Using systematic or local antibiotics that may influence tear producing

Elimianation Criteria

1. poor compliance
2. voluntary withdrawal
3. any other kind of situation that researchers consider not suitable for further study.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asian
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Tear cytokines levels | through study completion,an average of two weeks
  Comparision the tear cytokines （EGF, IL-17A, IL-1β, IL-8 and TNF-α）levels in different groups using using a Milliplex Map Kit (Human Th17 Magnetic Bead Panel, Millipore, Billerica, MA).

SECONDARY OUTCOMES:
Clinical correlations of the tear cytokines | through study completion,an average of two weeks
  Analysis of tear cytokines and clinical correlations by Spearman correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Hong Qi, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China